CLINICAL TRIAL: NCT05816161
Title: Comparison of The Effects of The Integrated Neuromuscular Inhibition Technique and Myofascial Release on Cervical Range of Motion and Dysfunction in Individuals With Nonspecific Cervical Pain
Brief Title: Integrated Neuromuscular Inhibition Technique and Myofascial Release on Cervical Range of Motion and Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall17/548
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Myofascial Trigger Point Pain
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Inhibition Technique (Experimental)
  Interventions: Diagnostic Test: Integrated Neuromuscular Inhibition Technique
- Myofascial Release (Other)
  Interventions: Diagnostic Test: Myofascial Release

INTERVENTIONS:
Diagnostic Test: Integrated Neuromuscular Inhibition Technique — Exercises
  Arms: Neuromuscular Inhibition Technique
Diagnostic Test: Myofascial Release — Exercises
  Arms: Myofascial Release

SUMMARY:
to findout the improvement by Integrated Neuromuscular Inhibition Technique and Myofascial Release on Cervical Range of Motion and Dysfunction

ELIGIBILITY:
Inclusion Criteria:

* ● Age between 25-40

  * Both males and females included
  * Participants suffering from recent cervical pain without any pathology.

Exclusion Criteria:

* ● Participants having cervical radiculopathy

  * Having recent trauma of the cervical spine
  * Non-cooperative subject

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Cervical Range of Motion measurement | 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudhary Muhammad Akram Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No